CLINICAL TRIAL: NCT01534403
Title: A Phase 2, Multicenter, Open-label, Long-term, Extension Study to Assess the Safety of Epratuzumab Treatment in Japanese Subjects With Systemic Lupus Erythematosus
Brief Title: Open Label Extension Study of Epratuzumab in Japanese Systemic Lupus Erythematosus (SLE) Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL0027
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Monoclonal antibody; B-cell immunotherapy; Epratuzumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epratuzumab 4x600 mg every 12 weeks Group (Experimental)
  Interventions: Biological: Epratuzumab

INTERVENTIONS:
Biological: Epratuzumab — Epratuzumab 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over eight 12-week treatment cycles (ie, Weeks 0, 1, 2, 3, 12, 13, 14, 15, 24, 25, 26, 27, 36, 37, 38, 39, 48, 49, 50, 51, 60, 61, 62, 63, 72, 73, 74, 75, 84, 85, 86, and 87)

SUMMARY:
The study is an open-labeled extension study to continue to assess the safety and tolerability of Epratuzumab in moderate to severe SLE subjects who have previously participated in SL0026 [NCT01449071] phase I/II trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the double-blind study SL0026 [NCT01449071] or terminated prematurely at Week 8 or later in SL0026 [NCT01449071] due to lack of efficacy
* Women of childbearing potential must agree to use an acceptable method of birth control/Written Informed Consent

Exclusion Criteria:

* Subjects with active, severe SLE disease activity which involves the renal system and active, severe, neuropsychiatric SLE, defined as any neuropsychiatric element scoring British Isles Lupus Assessment Group Index (BILAG) level A
* Subjects with concurrent relevant medical conditions like defined chronic infections or high risk of new significant infections
* Substance abuse or dependence
* Significant hematologic abnormalities
* History of malignant cancer
* Subjects with any other condition which, in the investigator's judgment, would make the subject unsuitable for inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting at least 1 Adverse Event (AE) during the Treatment Period (maximum 100 weeks) | up to Week 100
Change from Baseline in levels of total B Cells in the peripheral blood circulation at Week 96 | From Baseline (Week 0) to Week 96

SECONDARY OUTCOMES:
Change from Baseline in levels of Monocyte in the peripheral blood circulation at Week 96 | From Baseline (Week 0) to Week 96
Change from Baseline in levels of NK-Cells (Natural Killer-Cells) in the peripheral blood circulation at Week 96 | From Baseline (Week 0) to Week 96
Change from Baseline in levels of total T Cells in the peripheral blood circulation at Week 96 | From Baseline (Week 0) to Week 96
Epratuzumab plasma concentration at Week 96 | Week 96
Number of subjects reporting anti-Epratuzumab in plasma at Week 96 | Week 96

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (6):
- Japan (6):
  - 10, Fukuoka
  - 11, Fukuoka
  - 9, Fukuoka
  - 3, Kitakyushu
  - 1, Tokyo
  - 8, Tokyo